CLINICAL TRIAL: NCT01271387
Title: An Open-Label, Single-Dose, Parallel-Group Study to Compare the Pharmacokinetics of Tasimelteon With That in Matched Healthy Control Subjects
Brief Title: Pharmacokinetics of Tasimelteon in Subjects With Mild or Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VP-VEC-162-1105
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Hepatic Impairment
Keywords: Liver disease; pharmacokinetics
MeSH Terms: conditions — Liver Diseases | interventions — tasimelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: tasimelteon
- Mild Hepatic Impairment (Experimental)
  Interventions: Drug: tasimelteon
- Healthy Volunteers (Experimental)
  Interventions: Drug: tasimelteon

INTERVENTIONS:
Drug: tasimelteon — 20 mg tasimelteon capsules, PO single dose
  Other Names: VEC-162; BMS-214778

SUMMARY:
The purpose of this research study is to understand whether there is any difference in the amount of tasimelteon (including its breakdown products) in the blood in individuals with mild or moderate liver disease compared to individuals who have normal liver function.

DETAILED DESCRIPTION:
The study will employ an open-label, parallel-group design. Up to 32 subjects will be enrolled in 3 groups: Group 1 will consist of 8 subjects with mild hepatic impairment; Group 2 will consist of 8 subjects with moderate hepatic impairment; Group 3 will consist of up to 16 healthy subjects matched by gender, age, smoking status, and body mass index, to Groups 1 and/or 2. For each group, there will be a 21-day screening period, a baseline period, a single-dose treatment period with an on-site observation period of 36 hours, and a study completion evaluation conducted after the last PK blood sample is drawn. Each subject will receive a single 20-mg dose of tasimelteon, after which safety assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

* Ability and acceptance to provide written informed consent;
* Men or women between 18 - 75 years, inclusive;
* Subjects with Body Mass Index (BMI) of >18 and <35 kg/m2;
* Women of child-bearing potential must be using an acceptable method of birth control;
* Willing and able to comply with study requirements and restrictions;

Subjects with mild or moderate hepatic impairment:

* Stable hepatic impairment satisfying the criteria for Class A or B of the modified Child-Pugh classification documented by medical history;
* Subjects with Moderate hepatic impairment must also have either liver cirrhosis or physical signs consistent with a clinical diagnosis of liver cirrhosis
* Creatinine clearance greater than 50 mL/min

Healthy matched controls:

* Matched to subjects with hepatic impairment by gender, age, BMI, and smoking status
* Good health as determined by past medical history, physical examination, electrocardiogram, laboratory tests, vital signs and urinalysis;

Exclusion Criteria:

* Smokers unable or unwilling to limit consumption;
* Exposure to any investigational drug, including placebo, within 30 days of dosing;
* Blood Donation or loss of 400 mL or more within two months prior to dosing;
* Significant illness within the two weeks prior to dosing;
* History of autonomic dysfunction;
* History of acute or chronic bronchospastic disease, including asthma and chronic obstructive pulmonary disease, treated or not treated;
* A known hypersensitivity to tasimelteon or drugs similar to tasimelteon including melatonin;
* Pregnant or lactating females;
* History of drug or alcohol abuse within the 12 months prior to screening
* History of immunocompromise, including a positive HIV (ELISA and Western blot) test result;
* Any surgical or medical condition which might significantly alter the absorption, distribution or excretion of any drug;
* Clinically significant ECG abnormalities or vital sign abnormalities at screening or a history of unstable, severe, or clinically significant cardiovascular disease;

Subjects with mild or moderate hepatic impairment:

* Clinically significant abnormal findings, not consistent with clinical disease, upon physical examination, ECG, or laboratory evaluation;
* Current symptoms or past history (within the last 6 months) of encephalopathy;
* Severe ascites;
* Previous surgical porto-systemic shunt including transjugular intrahepatic portosystemic shunt (TIPS);
* Progressive liver disease within 4 weeks prior to screening.

Healthy matched controls:

* Use of any prescription medication within 1 month of dosing, and OTC medication within 14 days prior to dosing;
* History or presence of liver disease or liver injury;
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations and PK of tasimelteon | 36 hours
  To assess plasma concentrations and pharmacokinetics of tasimelteon in subjects with mild or moderate hepatic impairment compared to healthy subjects with normal hepatic function.

SECONDARY OUTCOMES:
Plasma concentrations and PK of tasimelteon metabolites | 36 hours
  To assess plasma concentrations and pharmacokinetics of tasimelteon metabolites in subjects with mild or moderate hepatic impairment compared to healthy subjects with normal hepatic function.
Safety | 36 hours
  To assess the safety and tolerability of a single 20-mg oral dose of tasimelteon.

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States